CLINICAL TRIAL: NCT00619450
Title: Three Dimensional C-Arm Computed Tomography of the Heart Chambers
Brief Title: Siemens 3-D C-Arm CT of the Heart Chambers
Acronym: DynaC-Arm
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-662
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; cardiac pacing; CAT scanner
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Other: 3D C-arm CT scan — The patient will be given an intravenous contrast dye and then hold their breath for 15 seconds while pictures are taken. The equipment used to take the pictures is like an arch that will rotate around the body. As the arch rotates, it will collect the pictures of the heart. These pictures will then be used to compute a three-dimensional image of the heart. The physicians will then continue with the planned procedure. The three-dimensional images will be reconstructed and available for the doctor to view during the case. The images will also be examined after the procedure by the physician.
  Other Names: DynaCT

SUMMARY:
The purpose of this study is to determine the optimal images of the heart structures which are used to guide AF ablation or BiVenticle and coronary vessels.

DETAILED DESCRIPTION:
'Atrial fibrillation (AF) and ventricular fibrillation are common sustained arrhythmias. The patient will be given an intravenous contrast dye and then hold their breath for 15 seconds while pictures are taken. The equipment used to take the pictures is like an arch that will rotate around the body. As the arch rotates, it will collect the pictures of the heart. These pictures will then be used to compute a three-dimensional image of the heart. The physicians will then continue with the planned procedure. The three-dimensional images will be reconstructed and available for the doctor to view during the case. The images will also be examined after the procedure by the physician.arrythmias of the heart, AF being the most common affecting over 5 million people world wide. While drugs are a first line therapy they can have significant side effects and are often not effective long term. AF ablation and cardiac resynchronization therapy (CRT) are emerging as a viable treatment options for many patients. Both treatments require a detailed knowledge of the anatomy of the heart so that instruments can be safely and accurately navigated within the heart to treat the condition. Detailed anatomical information is limited from 2D fluoroscopy and 3D information from preoperative computed tomography (CT) or electroanatomical mapping have inherent inaccuracies. 3D rotational angiography (C-arm CT) is a technology that will use the x-ray detector system in the EP room to create a 3D image of a section of the heart, such as the left atrium, in the EP treatment room at the onset of the ablation procedure. There are several potential advantages to this imaging technique; As the 3D image is created at the start of the procedure it is a better representation of the heart's anatomy at that time than data acquired days or weeks earlier; it may eliminate the need for a preoperative CT scan for many patients; C-arm CT exposes the patient to a lower radiation dose than a regular cardiac CT scan; and, as the scan is preformed in the EP room the physician has the opportunity to perform secondary scans should he suspect anything has changed during the procedure. The purpose of the research is to determine the optimal imaging protocol for the heart structures needed in cardiac procedures such as AF and CRT. The study will vary several imaging parameters such as contrast injection site, total contrast injected, injection rate, imaging system settings and data reconstruction parameters to determine the most appropriate protocol.'

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing EP diagnostic or therapeutic procedure
* Age > 18 years
* Male or Female
* Weight < 250 lbs
* Not pregnant - women without childbearing potential or women consenting to a pregnancy test
* Able to hold breath for a maximum of 15 seconds
* Sufficient kidney function to support a maximum of 200 cc of contrast in addition to whatever contrast will be given during the EP Procedure
* Creatinine < 1.7 AND cleared by physician prior to case
* Implantable foreign objects acceptable
* NSR or AF
* Patient must sign an informed consent

Exclusion Criteria:

* Patients should not have undergone a CT or CTA scan in the 24 hours prior to this study.
* Creatinine (GFR value) greater than 60

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female over age of 18 years and under 250 pounds undergoing a pulmonary vein isolation or implantation of cardiac pacemaker at the Cleveland Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To determine the optimal imaging protocol for the human heart structures which are used to guide AF ablation or biventricular pacing procedures, including the left atrium, left atrial appendage and pulmonary veins, left ventricle and coronary vessels. | 05/2008

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Cummings, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benndorf G, Strother CM, Claus B, Naeini R, Morsi H, Klucznik R, Mawad ME. Angiographic CT in cerebrovascular stenting. AJNR Am J Neuroradiol. 2005 Aug;26(7):1813-8. PMID 16091535
- [Background] Sze DY, Strobel N, Fahrig R, Moore T, Busque S, Frisoli JK. Transjugular intrahepatic portosystemic shunt creation in a polycystic liver facilitated by hybrid cross-sectional/angiographic imaging. J Vasc Interv Radiol. 2006 Apr;17(4):711-5. doi: 10.1097/01.RVI.0000208984.17697.58. PMID 16614155
- [Background] Lauritsch G, Boese J, Wigstrom L, Kemeth H, Fahrig R. Towards cardiac C-arm computed tomography. IEEE Trans Med Imaging. 2006 Jul;25(7):922-34. doi: 10.1109/tmi.2006.876166. PMID 16827492
- [Background] Moe GW, Canepa-Anson R, Howard RJ, Armstrong PW. Sequential changes in atrial pressures, dimensions, and plasma atrial natriuretic factor concentrations during volume loading in hemodynamically normal human subjects. J Lab Clin Med. 1991 Jun;117(6):528-34. PMID 1828490
- [Background] Welikovitch L, Lafreniere G, Burggraf GW, Sanfilippo AJ. Change in atrial volume following restoration of sinus rhythm in patients with atrial fibrillation: a prospective echocardiographic study. Can J Cardiol. 1994 Dec;10(10):993-6. PMID 7994668
- [Background] Zellerhoff M,Scholz B, Rührschopf E-P, Brunner T. "Low Contrast 3D-reconstruction from C-arm data", Proceeding of the SPIE, Vol. 5745, 146-655.
- [Background] Heran NS, Song JK, Namba K, Smith W, Niimi Y, Berenstein A. The utility of DynaCT in neuroendovascular procedures. AJNR Am J Neuroradiol. 2006 Feb;27(2):330-2. PMID 16484404
- [Background] Al-Ahmad A, Sandner-Porkristl D, Wigstrom L, Moore T, Boese J, Lauritsch G, Hsia H.H., Wang P.J., Fahrig R. Accuracy of Cardiac 3-D Image reconstruction of the Pulmonary Veins Using A Flat-panel C-arm CT System. Heart Rhythm Society Annual Scientific Sessions, May 2006, Boston, MA
- [Background] Nagel H.D. Radiation Exposure in Computed Tomography. European Coordinate Committee of the Radiological and Electromedical Industries (COCIR), Hamburg, 2000.
- [Background] Bongartz G, Golding S.J., Jurik A.G., et al. for the European Study Group. European guidelines on quality criteria for computed tomography. http://www.drs.dk/guidelines/ct/quality/mainindex.htm.
- [Background] Banckwitz R, Strobel N, Siemens Med AX, internal communication, April 27, 2006.